CLINICAL TRIAL: NCT06083636
Title: Improvement of Laboratory Diagnostics in Hypothyroid Patients Using Levothyroxine
Acronym: ANTICIPATE
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Annemieke Heijboer, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL81578.018.22
Record Dates: First submitted 2023-10-04; First posted 2023-10-16 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Hypothyroidism
Keywords: Hypothyroidism; Levothyroxine; Laboratory diagnostics; Free triiodothyronine; Central hypothyroidism
MeSH Terms: conditions — Hypothyroidism | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, plasma and serum samples are retained for 15 years as required for medical research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Hashimoto's hypothyroidism: Group of 100 patients with Hashimoto's hypothyroidism using levothyroxine
  Interventions: Other: Single extra blood draw and completion of single questionnaire
- Hypothyroidism after thyroidectomy after thyroid carcinoma: Group of 100 patients with hypothyroidism after thyroidectomy after thyroid carcinoma using levothyroxine
  Interventions: Other: Single extra blood draw and completion of single questionnaire
- Central hypothyroidism: Group of 100 patients with central hypothyroidism using levothyroxine
  Interventions: Other: Single extra blood draw and completion of single questionnaire
- Hypothyroidism during treatment for Graves' Disease: Group of 100 patients with hypothyroidism during treatment for Graves' Disease using levothyroxine
  Interventions: Other: Single extra blood draw and completion of single questionnaire
- Healthy controls: 100 healthy euthyroid controls
  Interventions: Other: Single blood draw and completion of single questionnaire

INTERVENTIONS:
Other: Single extra blood draw and completion of single questionnaire — Single blood draw of 3 tubes (20 mL) additional to regular blood draw will be performed. All participants will complete a single questionnaire that will be 5-10 minutes time-consuming.
  Groups: Central hypothyroidism; Hashimoto's hypothyroidism; Hypothyroidism after thyroidectomy after thyroid carcinoma; Hypothyroidism during treatment for Graves' Disease
Other: Single blood draw and completion of single questionnaire — Single blood draw of 3 tubes (20 mL) will be performed. All participants will complete a single questionnaire that will be 5-10 minutes time-consuming.
  Groups: Healthy controls

SUMMARY:
Hypothyroidism is a thyroid disorder and one of the most common endocrine disorders. Hypothyroidism can have multiple causes; most patients suffer from primary autoimmune hypothyroidism (Hashimoto's disease), but also central hypothyroidism, hypothyroidism after total thyroidectomy due to thyroid carcinoma, or hypothyroidism due to therapy of Graves' disease occur. Most patients with hypothyroidism are treated with levothyroxine (L-T4) to supplement the lack of thyroxine (T4) produced by their own thyroid. Serum thyroid-stimulating hormone (TSH) and/or free T4 (fT4) are currently measured to assess the efficacy of this therapy and to establish euthyroidism. It is known that fT4 concentrations in patients using L-T4 can be above the upper limit of the reference interval, while their TSH is not (completely) suppressed. This raises the question whether fT4 is an accurate reflection of thyroid hormone status in patients using L-T4. TSH is considered a reliable parameter of thyroid hormone status; however, TSH cannot be used to assess thyroid function in specific hypothyroid patient groups (e.g. central hypothyroidism). Free triiodothyronine (fT3), the active thyroid hormone, has been suggested to be an interesting alternative of fT4 to assess thyroid function. Previously, the methods to measure fT3 were not that robust; however, methods to determine fT3 have been improved, are currently reliable and not susceptible to changes due to L-T4 intake. In addition, the fT3/fT4 ratio is thought to be an interesting candidate in assessing thyroid hormone status as well. The aim of this study is to improve laboratory diagnostics of thyroid hormone status in patients with hypothyroidism receiving L-T4 in whom TSH cannot be used as a reflection of thyroid hormone status. We will primarily investigate the additional already available laboratory tests fT3 and fT3/fT4 ratio. We hypothesize that treated hypothyroid participants who are assumed euthyroid based on TSH (e.g. patients with Hashimoto's hypothyroidism) but have fT4 concentrations above the upper reference limit will more often have a fT3 level or a fT3/fT4 ratio within the reference interval. Concentrations of alternative markers in healthy controls and patients with Hashimoto's hypothyroidism with 'normal' TSH concentrations can, thus, be used to predict thyroid hormone status in patients using L-T4 in whom TSH cannot be used to assess thyroid hormone status.

DETAILED DESCRIPTION:
Hypothyroidism is a thyroid disorder and one of the most common endocrine disorders. Hypothyroid patients have a thyroid hormone deficiency characterized by a shortage of thyroid hormone (TH) in the circulation and at the organ level and are normally treated with a synthetic form of thyroid hormone (L-T4 or levothyroxine). Thyroxine (T4) is a prohormone, produced by the thyroid gland and converted into the active hormone triiodothyronine (T3) in peripheral tissues. A minor percentage (20%) of circulating T3 is directly produced by the thyroid gland. Although L-T4 treatment accounts for all patients with hypothyroidism, the pathogenesis of hypothyroidism differs. Most patients suffer from primary hypothyroidism (Hashimoto's disease), which is an auto-immune disorder, but also central hypothyroidism, hypothyroidism after total thyroidectomy due to thyroid carcinoma or hypothyroidism due to therapy of Graves' disease are commonly seen.

Currently, thyroid-stimulating hormone (TSH) and/or free T4 (fT4) are measured in serum to monitor the treatment efficacy of L-T4. TSH is produced by the pituitary to stimulate the production of thyroid hormones by the thyroid gland and due to the negative feedback loop considered as a good reflection of thyroid hormone status. Target concentrations of TSH and fT4 differ depending on the cause of hypothyroidism. In patients with Hashimoto's hypothyroidism, TSH concentrations are measured to monitor treatment and TSH levels within the reference intervals are pursued. TSH is measured to monitor treatment in patients with hypothyroidism after total thyroidectomy due to thyroid carcinoma as well, although a suppressed TSH is warranted in this group. The extent of TSH suppression is determined based on the type and stage of the carcinoma. In patients who are hypothyroid due to therapy of Graves' disease, other target values apply. Patients who are just diagnosed with Graves' disease start with thyroid suppressive therapy together with thyroid hormone supplementation (L-T4) and show a prolonged suppressed TSH; therefore, fT4 is initially used to monitor therapy. TSH is used to monitor treatment again when TSH starts to normalize. Nevertheless, TSH shall always be slightly suppressed due to the TSH receptor antibodies produced during Graves' disease, which means fT4 concentration is still taken into account during follow-up. Finally, it is not possible to monitor treatment by using TSH concentrations in patients with central hypothyroidism, which means fT4 concentrations are leading in this group. In conclusion, TSH cannot always be used to assess thyroid function in which cases fT4 is assessed as well.

It is known that patients using L-T4 can show a combination of fT4 values above the upper reference limit and non-suppressed or only slightly suppressed TSH levels. The most likely explanation for this is twofold. First, thyroid hormones are supplemented by L-T4, which only replaces T4, whereas the production of the active thyroid hormone T3 by the thyroid gland is lacking and the patients depend on peripheral conversion of T4. Literature showed that these patients need a higher L-T4 dosage to obtain a normal, or even somewhat lower, concentration of T3. TSH is regulated by changes in T3 rather than T4, clarifying the lack of pituitary feedback to increased fT4 concentrations if fT3 concentrations are not increased simultaneously. Second, previous studies showed that fT4 levels peak two until four hours after L-T4 intake and gradually decline until the next dosage is taken. Sometimes, this peak increases above the upper limit of the reference interval. This pattern is not seen for TSH levels. Looking at aforementioned outcomes, it seems that fT4 levels are higher in patients using L-T4 compared to healthy controls, thus not reflecting thyroid hormone status adequately.

In clinical practice, the largest group of hypothyroid patients are monitored by measuring TSH as mentioned above. Therefore, these high fT4 levels will only rarely cause problems. However, these high fT4 levels can have treatment consequences in patient groups wherein therapy is monitored via fT4 levels (e.g. central hypothyroidism), which could lead to unwarranted dose adjustments (leading to a too low dose of L-T4).

Free T3 (fT3) concentrations can be measured but are used only rarely in clinical practice. Previously, the fT3 measurement using immunoassay techniques was troublesome and, therefore, considered as unreliable. However, the quality of the currently used immunoassay has been substantially improved resulting in the availability of reliable fT3 immunoassays. Furthermore, in contrast to fT4, fT3 is not subject to change after L-T4 intake. Consequently, fT3 might be an interesting parameter to assess thyroid hormone status in L-T4 users along with TSH. In addition, literature suggested that the ratio between fT3 and fT4 might be worthwhile investigating as an indicator of peripheral conversion. The fT3/fT4 ratio is thought to be lower in L-T4 users compared to euthyroid controls and could, therefore, be used to evaluate to what extent T4 is converted to T3. A decline might represent insufficient availability of thyroid hormone throughout the body.

Thyroid hormone markers as total T4 (TT4) and total T3 (TT3) were used as thyroid hormone parameters before the free fractions of both thyroid hormones (fT4 and fT3) could be used. They lost ground as traditional thyroid hormone biomarkers but still provide relevant information about general thyroid hormone status. Degradation of T4 results in the formation of reversed T3 (rT3). This thyroid hormone biomarker can be measured in serum and has already proven to be of significance in the diagnosis of non-thyroidal illness syndrome (NTIS). However, it might also be useful as biomarker in patients using L-T4. Furthermore, several biomarkers have been proposed to evaluate tissue thyroid hormone status and to provide a better insight into thyroid hormone status in peripheral tissues, such as sex-hormone binding globulin (SHBG), acylcarnitines and several amino acids. Although these biomarkers are not directly proposed as better suitable biomarkers than fT4 in patients using L-T4, it will be interesting to assess their contribution and relevance in this specific patient group. Deiodinases (DIO1, DIO2 and DIO3) greatly contribute to the conversion of inactive T4 to active T3 and to the degradation of thyroid hormones. DIO polymorphisms are common in the general population and might influence the treatment efficacy of certain patients using L-T4 and could, thus, be interesting to take into account.

As previously mentioned, some biomarkers indicating thyroid hormone status show a shifted normal distribution compared to healthy controls. To assess to what extent other biomarkers contribute to indicate thyroid status, it is necessary to know what the normal distributions of these biomarkers are in the healthy population. After that, results in patient groups using L-T4 can be assessed and compared to results of healthy controls. Therefore, healthy controls must be included to obtain valid results.

The aim of this study is to investigate whether a variety of additional markers can improve laboratory diagnostics in patients with hypothyroidism receiving L-T4 in whom TSH cannot be used as a reflection of thyroid hormone status (e.g. central hypothyroidism). Alternatives could be fT3 and the derived fT3/fT4 ratio but TT4, TT3, rT3, SHBG, acylcarnitines and several amino acids might be interesting parameters as well. We hypothesize that treated hypothyroid participants who are assumed euthyroid based on TSH (e.g. patients with Hashimoto's hypothyroidism) but have fT4 concentrations above the upper reference limit will more often have a fT3 level or a fT3/fT4 ratio within the reference interval. TSH is considered to reflect thyroid hormone status reliably. Concentrations of alternative markers in healthy controls and patients with Hashimoto's hypothyroidism with 'normal' TSH concentrations can, thus, be used to predict thyroid hormone status in patients using L-T4 in whom TSH cannot be used to assess thyroid hormone status. Therefore, outcomes of this study will particularly benefit the follow-up of patients with central hypothyroidism in whom TSH cannot be used to monitor thyroid hormone status.

After informed consent is provided, participation to the study entails a single blood draw (3 tubes, 20 mL) and a single questionnaire (ThyPRO-39), the study is thus of cross-sectional design. Blood draw from hypothyroid patients using L-T4 is performed at the same time as regular blood draw. Therefore, no extra blood draw is necessary. Healthy controls will undergo one blood withdrawal. All data are stored pseudo-anonymously.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a hypothyroid subject must meet all of the following criteria:

* Ability to provide informed consent
* Ability to speak and understand Dutch or English
* Intake of a stable dosage of levothyroxine, meaning the dosage of levothyroxine must not be changed during the appointment at the outpatient clinic
* Diagnosis of one these forms of hypothyroidism

  * Patients with primary hypothyroidism: euthyroid based on TSH according to physician
  * Patients with hypothyroidism after a total thyroidectomy due to thyroid carcinoma (therefore athyroid): on target TSH according to physician (target TSH depending on stage/severity of carcinoma)
  * Patients using L-T4 due to therapy of Graves' disease: euthyroid based on TSH according to physician (TSH cannot be suppressed, namely TSH within reference interval of 0,5-5,0 mU/L)
  * Patients with central hypothyroidism: euthyroid based on fT4 according to physician (common is fT4 in the upper limit, reference interval is 12-22 pmol/L)

In order to be eligible to participate in this study, a healthy control subject must meet all of the following criteria:

* Ability to provide informed consent;
* Ability to speak and understand Dutch or English
* Consider themselves healthy

Exclusion Criteria:

A potential hypothyroid subject who meets any of the following criteria will be excluded from participation in this study:

* Not euthyroid according to physician
* Pregnancy
* Patients using L-T4 due to therapy of Graves' disease: if TSH is still suppressed
* Any of the following medication

  * Liothyronine (Cytomel)
  * Iodide
  * Oral contraceptives
  * Active treatment of malignancy (other than thyroid carcinoma)

A potential healthy control subject who meets any of the following criteria will be excluded from participation in this study:

* Pregnancy
* Any of the following medication

  * Thyroid medication (a.o. levothyroxine, thiamazol, PTU)
  * Lithium
  * Amiodarone
  * Propranolol
  * Iodide
  * Glucocorticoids
  * Oral contraceptives
  * Heparin
  * Growth hormone
  * Active treatment of malignancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with hypothyroidism using levothyroxine (L-T4) attending the outpatient clinic of Amsterdam UMC will be included. Healthy euthyroid controls will be recruited amongst employees of Amsterdam UMC.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
TSH concentration | Single measurement in cross-sectional design during the study period, which is approximately 4 years
  Laboratory measurement
fT4 concentration | Single measurement in cross-sectional design during the study period, which is approximately 4 years
  Laboratory measurement
fT3 concentration | Single measurement in cross-sectional design during the study period, which is approximately 4 years
  Laboratory measurement
fT3/fT4 ratio | One-time determination in cross-sectional design during the study period, which is approximately 4 years
  Ratio derived from abovementioned laboratory measurements

SECONDARY OUTCOMES:
TT4 concentration | Single measurement in cross-sectional design during the study period, which is approximately 4 years
  Laboratory measurement
TT3 concentration | Single measurement in cross-sectional design during the study period, which is approximately 4 years
  Laboratory measurement
rT3 concentration | Single measurement in cross-sectional design during the study period, which is approximately 4 years
  Laboratory measurement
SHBG | Single measurement in cross-sectional design during the study period, which is approximately 4 years
  Laboratory measurement
Acylcarnitine(s) (profile) | Single measurement in cross-sectional design during the study period, which is approximately 4 years
  Laboratory measurement
Amino acids | Single measurement in cross-sectional design during the study period, which is approximately 4 years
  Laboratory measurement

OTHER OUTCOMES:
ThyPRO-39 | One-time completion around time of laboratory measurement during the study period, which is approximately 4 years
  Questionnaire
DIO polymophisms | Single measurement in cross-sectional design during the study period, which is approximately 4 years
  Laboratory measurement
Sex | One-time completion around time of laboratory measurement during the study period, which is approximately 4 years
  Questionnaire; patient characteristics
Age | One-time completion around time of laboratory measurement during the study period, which is approximately 4 years
  Questionnaire; patient characteristics
Smoking status | One-time completion around time of laboratory measurement during the study period, which is approximately 4 years
  Questionnaire; patient characteristics
Co-medication | One-time completion around time of laboratory measurement during the study period, which is approximately 4 years
  Questionnaire; patient characteristics
Cause of hypothyroidism | One-time completion around time of laboratory measurement during the study period, which is approximately 4 years
  Questionnaire; patient characteristics
Time of L-T4 intake | One-time completion around time of laboratory measurement during the study period, which is approximately 4 years
  Questionnaire; patient characteristics
Dosage of L-T4 | One-time completion around time of laboratory measurement during the study period, which is approximately 4 years
  Questionnaire; patient characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Annemieke C Heijboer, Prof. dr., Principal Investigator — Amsterdam UMC, VU Amsterdam and UvA, Endocrine Laboratory, Department of Laboratory Medicine
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garmendia Madariaga A, Santos Palacios S, Guillen-Grima F, Galofre JC. The incidence and prevalence of thyroid dysfunction in Europe: a meta-analysis. J Clin Endocrinol Metab. 2014 Mar;99(3):923-31. doi: 10.1210/jc.2013-2409. Epub 2014 Jan 1. PMID 24423323
- [Background] Gullo D, Latina A, Frasca F, Le Moli R, Pellegriti G, Vigneri R. Levothyroxine monotherapy cannot guarantee euthyroidism in all athyreotic patients. PLoS One. 2011;6(8):e22552. doi: 10.1371/journal.pone.0022552. Epub 2011 Aug 1. PMID 21829633
- [Background] Woeber KA. Levothyroxine therapy and serum free thyroxine and free triiodothyronine concentrations. J Endocrinol Invest. 2002 Feb;25(2):106-9. doi: 10.1007/BF03343972. PMID 11929079
- [Background] Peterson SJ, McAninch EA, Bianco AC. Is a Normal TSH Synonymous With "Euthyroidism" in Levothyroxine Monotherapy? J Clin Endocrinol Metab. 2016 Dec;101(12):4964-4973. doi: 10.1210/jc.2016-2660. Epub 2016 Oct 4. PMID 27700539
- [Background] Deam DR, Campbell DG, Ratnaike S. Effect of oral intake of thyroxine on results of thyroid function tests in patients receiving thyroid replacement therapy. Med J Aust. 1983 Oct 15;2(8):374-6. doi: 10.5694/j.1326-5377.1983.tb122530.x. PMID 6621483
- [Background] Browning MC, Bennet WM, Kirkaldy AJ, Jung RT. Intra-individual variation of thyroxin, triiodothyronine, and thyrotropin in treated hypothyroid patients: implications for monitoring replacement therapy. Clin Chem. 1988 Apr;34(4):696-9. PMID 3359603
- [Background] Saravanan P, Siddique H, Simmons DJ, Greenwood R, Dayan CM. Twenty-four hour hormone profiles of TSH, Free T3 and free T4 in hypothyroid patients on combined T3/T4 therapy. Exp Clin Endocrinol Diabetes. 2007 Apr;115(4):261-7. doi: 10.1055/s-2007-973071. PMID 17479444
- [Background] Soppi E, Irjala K, Kaihola HL, Viikari J. Acute effect of exogenous thyroxine dose on serum thyroxine and thyrotrophin levels in treated hypothyroid patients. Scand J Clin Lab Invest. 1984 Jun;44(4):353-6. doi: 10.3109/00365518409083819. PMID 6463564
- [Background] Czernichow P, Wolf B, Fermanian J, Pomarede R, Rappaport R. Twenty-four hour variations of thyroid hormones and thyrotrophin concentrations in hypothyroid infants treated with L-thyroxine. Clin Endocrinol (Oxf). 1984 Oct;21(4):393-7. doi: 10.1111/j.1365-2265.1984.tb03226.x. PMID 6509783
- [Background] Wennlund A. Variation in serum levels of T3, T4, FT4 and TSH during thyroxine replacement therapy. Acta Endocrinol (Copenh). 1986 Sep;113(1):47-9. doi: 10.1530/acta.0.1130047. PMID 3766048
- [Background] Symons RG, Murphy LJ. Acute changes in thyroid function tests following ingestion of thyroxine. Clin Endocrinol (Oxf). 1983 Oct;19(4):539-46. doi: 10.1111/j.1365-2265.1983.tb00029.x. PMID 6627702
- [Background] Dong BJ, Hauck WW, Gambertoglio JG, Gee L, White JR, Bubp JL, Greenspan FS. Bioequivalence of generic and brand-name levothyroxine products in the treatment of hypothyroidism. JAMA. 1997 Apr 16;277(15):1205-13. PMID 9103344
- [Background] Ain KB, Pucino F, Shiver TM, Banks SM. Thyroid hormone levels affected by time of blood sampling in thyroxine-treated patients. Thyroid. 1993 Summer;3(2):81-5. doi: 10.1089/thy.1993.3.81. PMID 8369656
- [Background] Hoermann R, Midgley JEM, Dietrich JW, Larisch R. Dual control of pituitary thyroid stimulating hormone secretion by thyroxine and triiodothyronine in athyreotic patients. Ther Adv Endocrinol Metab. 2017 Jun;8(6):83-95. doi: 10.1177/2042018817716401. Epub 2017 Jul 13. PMID 28794850
- [Background] Hoermann R, Midgley JE, Larisch R, Dietrich JW. Is pituitary TSH an adequate measure of thyroid hormone-controlled homoeostasis during thyroxine treatment? Eur J Endocrinol. 2013 Jan 17;168(2):271-80. doi: 10.1530/EJE-12-0819. Print 2013 Feb. PMID 23184912
- [Background] Strich D, Chay C, Karavani G, Edri S, Gillis D. Levothyroxine Therapy Achieves Physiological FT3/FT4 Ratios at Higher than Normal TSH Levels: A Novel Justification for T3 Supplementation? Horm Metab Res. 2018 Nov;50(11):827-831. doi: 10.1055/a-0751-0498. Epub 2018 Nov 5. PMID 30396211
- [Background] Iwayama H, Sugahara K, Nakano M, Fukayama M, Okumura A. Measurement of reverse triiodothyronine levels using liquid chromatography-tandem mass spectrometry in the serum of 89 outpatients. Medical Mass Spectrometry. 2017;1(1):10-3.
- [Background] Docter R, Krenning EP, de Jong M, Hennemann G. The sick euthyroid syndrome: changes in thyroid hormone serum parameters and hormone metabolism. Clin Endocrinol (Oxf). 1993 Nov;39(5):499-518. doi: 10.1111/j.1365-2265.1993.tb02401.x. No abstract available. PMID 8252737
- [Background] Dumoulin SC, Perret BP, Bennet AP, Caron PJ. Opposite effects of thyroid hormones on binding proteins for steroid hormones (sex hormone-binding globulin and corticosteroid-binding globulin) in humans. Eur J Endocrinol. 1995 May;132(5):594-8. doi: 10.1530/eje.0.1320594. PMID 7749500
- [Background] Harrison SA, Bashir MR, Guy CD, Zhou R, Moylan CA, Frias JP, Alkhouri N, Bansal MB, Baum S, Neuschwander-Tetri BA, Taub R, Moussa SE. Resmetirom (MGL-3196) for the treatment of non-alcoholic steatohepatitis: a multicentre, randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2019 Nov 30;394(10213):2012-2024. doi: 10.1016/S0140-6736(19)32517-6. Epub 2019 Nov 11. PMID 31727409
- [Background] Chng CL, Lim AY, Tan HC, Kovalik JP, Tham KW, Bee YM, Lim W, Acharyya S, Lai OF, Chong MF, Yen PM. Physiological and Metabolic Changes During the Transition from Hyperthyroidism to Euthyroidism in Graves' Disease. Thyroid. 2016 Oct;26(10):1422-1430. doi: 10.1089/thy.2015.0602. Epub 2016 Sep 7. PMID 27465032
- [Background] Al-Majdoub M, Lantz M, Spegel P. Treatment of Swedish Patients with Graves' Hyperthyroidism Is Associated with Changes in Acylcarnitine Levels. Thyroid. 2017 Sep;27(9):1109-1117. doi: 10.1089/thy.2017.0218. Epub 2017 Aug 18. PMID 28699427
- [Background] Castagna MG, Dentice M, Cantara S, Ambrosio R, Maino F, Porcelli T, Marzocchi C, Garbi C, Pacini F, Salvatore D. DIO2 Thr92Ala Reduces Deiodinase-2 Activity and Serum-T3 Levels in Thyroid-Deficient Patients. J Clin Endocrinol Metab. 2017 May 1;102(5):1623-1630. doi: 10.1210/jc.2016-2587. PMID 28324063
- [Background] Jo S, Fonseca TL, Bocco BMLC, Fernandes GW, McAninch EA, Bolin AP, Da Conceicao RR, Werneck-de-Castro JP, Ignacio DL, Egri P, Nemeth D, Fekete C, Bernardi MM, Leitch VD, Mannan NS, Curry KF, Butterfield NC, Bassett JHD, Williams GR, Gereben B, Ribeiro MO, Bianco AC. Type 2 deiodinase polymorphism causes ER stress and hypothyroidism in the brain. J Clin Invest. 2019 Jan 2;129(1):230-245. doi: 10.1172/JCI123176. Epub 2018 Dec 3. PMID 30352046